CLINICAL TRIAL: NCT05270876
Title: A Feasibility, Prospective, Repeated-measures Investigation to Investigate Innovations in Clinical Care in Adult and Paediatric Recipients Implanted With CE Approved Nucleus Cochlear Implants: an Umbrella Investigation
Brief Title: Innovations in Clinical Care of CE Approved Nucleus Cochlear Implant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AI5763
Record Dates: First submitted 2021-09-28; First posted 2022-03-08 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-12

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Cochlear Implants; Diagnosis; Weights and Measures

STUDY DESIGN:
Intervention Model Description: Interrupted time series
Masking Description: Participants were masked to which fitting method they had at any point in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study cohort (Other): Recipients of cochlear implant or suitable for implantation Interrupted time series: recipients received standard and novel fitting method
  Interventions: Device: Cochlear Implant and sound processor device fitting paradigm or diagnostic/measurement technique

INTERVENTIONS:
Device: Cochlear Implant and sound processor device fitting paradigm or diagnostic/measurement technique — The investigational device will be a new device fitting paradigm or diagnostic/measurement technique implemented for use with the commercially available sound processor and implant.

SUMMARY:
This study is to evaluate new approaches to device fitting and diagnostics for cochlear implant users. The evaluation can be performed in the laboratory in an acute session or in real world environments with take-home device use to further validate their benefits. Each feature will be tested in a sub-study specific to that hearing care model. On average, each sub-study is expected to include approximately 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Users of a CE approved Nucleus cochlear implant, resulting in open set speech understanding
* At least three months of experience with the cochlear implant.
* Older than 18 years when entering the study.
* Subject is fluent speaker in the language used for assessments.
* Open set speech understanding sufficient to complete the study protocol as judged by the investigator.
* Willing and able to provide written informed consent

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the investigator.
* Additional health factors, known to the investigator, that would prevent or restrict participation in the audiological evaluations.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organizations or contractors engaged by Cochlear for the purposes of this investigation.
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (2):
  - HEARnet Clinical Studies - The University of Melbourne, Carlton, Victoria
  - Cochlear Ltd. Melbourne, East Melbourne, Victoria
- Belgium (3):
  - AZ Sint-Jan Brugge-Oostende AV, Bruges, België
  - Sint-Augustinus Antwerpen, Wilrijk, België
  - Cochlear Technology Centre Belgium, Mechelen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Cohort: Recipients of cochlear implant or suitable for implantation
  Recipients received standard and novel fitting methods during the study
Period: Overall Study
Arm/Group | Study Cohort
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Cohort
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 66.5 [26 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Average period of CI experience [Mean (Full Range); unit: years] | 5.3 [0.25 to 13]
Device type [Count of Participants; unit: Participants]
  CI532 | 11
  CI632 | 3
  CI512 | 3
  CI612 | 1
  CI24RE(CS) | 1
  CI24RE(CA) | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference Between Standard and Novel Fitting Method for Monosyllabic Word Scores in Quiet
Description: The difference between mean CNC scores (reported as percentage of correct answers) in quiet between the standard and novel fitting method
Time Frame: 0 to 4 weeks after fitting
Population: All study recipients received the standard and novel fitting methods at different timepoints of the study.
Measure: Mean (95% Confidence Interval); unit: difference in percentage correct answers
Groups:
- Study Cohort: Recipients of cochlear implant or suitable for implantation
Arm/Group | Study Cohort
Number analyzed (Participants) | 20
difference in percentage correct answers | 3.8 [-1.041 to 8.641]

ADVERSE EVENTS:
Time Frame: 3 weeks
Description: Subjects were monitored over the study duration which was approximately 3 weeks.
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study Cohort (N=20)
Headache (General disorders) | 2
Discomfort (General disorders) | 3
Dizziness (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT05270876/Prot_SAP_001.pdf